CLINICAL TRIAL: NCT03348553
Title: Bioavailability of Major Compounds of a Vegan Fatty-acid Nutraceutical and Its Effect on the Lipid Profile in Individuals With Suboptimal Serum-lipid Values
Brief Title: Juice Plus+OMEGA Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Green Beat (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Lamprecht Manfred PhD, PhD, Sponsor Investigator, Green Beat
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 29-525ex16/17
Record Dates: First submitted 2017-11-03; First posted 2017-11-21 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Healthy
Keywords: Omega-fatty-acids; Absorption; Bioavailability; Fruit & Vegetable concentrate; Lipid Metabolism
MeSH Terms: interventions — Control Groups; omega-(4-iodophenyl)pentadecanoic acid

STUDY DESIGN:
Intervention Model Description: subjects are randomised into one of 4 intervention groups (control group (CG; consumption of 2 capsules of JP+® Omega Blend/d (Ω2); consumption of 4 capsules JP+® Omega Blend/d (Ω4); consumption of 2 capsules JP+® Omega Blend + Juice Plus+® fruit, vegetable and berry juice concentrate with 2 capsules each /d (Ω2+OGV)). Subjects allocated to Ω2 and Ω4 will receive the herbal fatty acid nutraceutical in the 4-month long study period (intervention phase), subjects allocated to Ω2+OGV will additionally receive the fruit, vegetable and berry juice concentrate. The control group will refrain from using any supplements over the course of this period and will maintain their usual eating habits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (Sham Comparator): 20 subjects do not receive any supplementation
  Interventions: Dietary Supplement: control group
- Omega2 (Active Comparator): 20 subjects receive an Omega-Fatty-acid Nutratceutical
  Interventions: Dietary Supplement: Omega2
- Omega4 (Active Comparator): 20 subjects receive an Omega-Fatty-acid Nutraceutical
  Interventions: Dietary Supplement: Omega4
- Omega2+OGV (Active Comparator): 20 subjects receive an Omega-Fatty-acid Nutraceutical + encapsulated fruit, vegetable and berry-juice concentrate
  Interventions: Dietary Supplement: Omega2+OGV

INTERVENTIONS:
Dietary Supplement: control group — no supplements given for 16 weeks, after 4 week washout of all supplements and dietetic products
  Arms: control group
Dietary Supplement: Omega2 — 2 capsules of JP+® Omega/d for 16 weeks, after 4 week washout of all supplements and dietetic products
  Arms: Omega2
Dietary Supplement: Omega4 — 4 capsules of JP+® Omega/d for 16 weeks, after 4 week washout of all supplements and dietetic products
  Arms: Omega4
Dietary Supplement: Omega2+OGV — 2 capsules of JP+® Omega/d plus 2 capsules each of an encapsulated fruit, vegetable and berry-juice concentrate (6 capsules) for 16 weeks, after 4 week washout of all supplements and dietetic products
  Arms: Omega2+OGV

SUMMARY:
In this randomized, controlled clinical study firstly the bioavailability of fatty acids and micronutrients of JP+® Omega Blend will be analysed. Secondly, the effect of the constituents contained in the nutraceuticals on blood lipid values will be determined. Thirdly, it will be examined, whether a dose-dependent effect of the supplementation of JP+® Omega Blend exists. Fourthly, the effect of a combined consumption of JP+® Omega Blend and Juice Plus+® Orchard, Garden and Vineyard blend (JP+® OGV) is investigated.

DETAILED DESCRIPTION:
In this randomized, controlled clinical study firstly the bioavailability of fatty acids and micronutrients of JP+Omega Blend will be analysed. Secondly, the effect of the constituents contained in the nutraceuticals on blood lipid values will be determined. Thirdly, it will be examined, whether a dose-dependent effect of the supplementation of JP+ Omega Blend exists. Fourthly, the effect of a combined consumption of JP+ Omega Blend and Juice Plus+® Orchard, Garden and Vineyard blend (JP+ OGV) is investigated.

RESEARCH QUESTIONS:

* To which extend will the ω-3-fatty acids, as well as certain micronutrients, such as carotenoids and tocopherols contained in the herbal fatty acid nutraceutical JP+® Omega Blend be resorbed?
* Are the ω-3 fatty acids bioavailable by increasing ω-3-index?
* Does a 4-month long supplementation with a plant-based herbal fatty acid nutraceutical (JP+ Omega Blend) exert a positive effect on lipid metabolism in subjects with suboptimal serum-lipid values?
* Does a dose-dependent effect on lipid profile exist in the subjects through supplementation of JP+ Omega Blend?
* Does the supply of JP+ Omega Blend combined with JP+® OGV exert different or additional effects on bioavailability and lipid metabolism in subjects with suboptimal serum-lipid values?

HYPOTHESES

1. We hypothesise that the ω-3-fatty acids of JP+ Omega Blend will be absorbed in significant amounts in a dose-dependent manner and have a good bioavailability.
2. We pursue the hypothesis, that the supplementation of JP+Omega Blend - at different dosage or combined with the consumption of JP+ OGV - will cause a positive effect on lipid metabolism in subjects with suboptimal serum-lipid values.
3. Additionally, we hypothesise that carotenoids and tocopherols (="micronutrients") contained in Juice Plus+Omega Blend will be absorbed.

The "null-hypotheses" are in detail:

1. The ω-3-fatty acids, contained in JP+Omega Blend, are not significantly absorbed.
2. The ω-3-fatty acids, contained in JP+Omega Blend, show no bioavailability or no increase in erythrocyte ω-3-index, respectively.
3. The supplementation of JP+ Omega Blend in different dosages and combined with the supplementation of JP+ OGV has no (additional) effect on lipid profile and /or metabolism in subjects with suboptimal serum lipid values.
4. The carotenoids and tocopherols contained in JP+®Omega Blend are not absorbed to a significant extent.

ENDPOINTS

• Primary endpoint: Ω-3-index = bioavailability of ω-3-fatty acids

* Secondary endpoint: lipid profile
* Tertiary endpoint: absorption of micronutrients

AIMS

This randomised, controlled, clinical study evaluates:

1. The bioavailability of omega-3 fatty acids of a herbal fatty acid nutraceutical (JP+® Omega Blend) after two and four months supplementation.
2. The effects of a 4-month long supplementation period of JP Omega-Blend in different dosages or combined with a fruit, vegetable and berry juice concentrate (JP+® selection of fruit, vegetables, and berries) on bioavailability and lipid metabolism in subjects with suboptimal serum lipid values.

   MERITS

   - The data acquired within this project will provide scientifically sound information about absorption and bioavailability of ω-3-fatty acids contained in the herbal nutraceutical Juice Plus+ Omega Blend.

   - The results of this project will provide information about the effect of the supplementation of a purely herbal fatty acid product on lipid metabolism in subjects with suboptimal serum lipid values.

   - Data of this study will provide information about a possible dose-dependent effect of JP+Omega Blend supplementation and an effect of the combined supplementation of JP+Omega Blend and JP+ OGV on lipid metabolism and micronutrient absorption in subjects with suboptimal serum lipid values.

   METHODS/STUDY DESIGN

   • Study design: This clinical study is a randomized, controlled study with a parallel-group design.

   The recruitment phase of the study starts with initial telephone interviews of potential subjects about inclusion and exclusion criteria for pre-selection. Special focus will lie on the determination of any intake of nutritional supplements including antioxidants, supplements with relevant effects on redox biology, omega-3 fatty acids and various plant extracts and concentrates. If a supplementation with the just mentioned substances is conducted, a wash-out phase of at least 4 weeks has to be implemented before the pre-screening period. The pre-screening aims to further evaluate inclusion and exclusion criteria of the subjects and also focuses on the measurement of ω-3 indices and blood pressure.

   If inclusion criteria are met and written informed consent is given, subjects are randomised into one of 4 intervention groups (control group (CG; consumption of 2 capsules of JP+ Omega Blend/d (Ω2); consumption of 4 capsules JP+ Omega Blend/d (Ω4); consumption of 2 capsules JP+ Omega Blend + Juice Plus+ Obst-, Gemüse- und Beerensaftkonzentrat with 2 capsules each /d (Ω2+OGV)). Subjects allocated to Ω2 and Ω4 will receive the herbal fatty acid nutraceutical in the 4-month long study period (intervention phase), subjects allocated to Ω2+OGV will additionally receive the fruit, vegetable and berry juice concentrate. The control group will refrain from using any supplements over the course of this period and will maintain their usual eating habits.

   Subjects are asked to complete an at least 4-week long wash-out phase, before attending the baseline-visit. The consumption of foods, as well as medication and supplements, which could influence the study outcome, will be suspended (see section "nutrition").

   The measurements and examinations with eligible subjects will be conducted within the scope of the study visits at baseline, after 2 (midpoint) and after 4 months (end of study; endpoint).

   • Subjects The subjects of this study comprise 80 healthy men and women with suboptimal serum lipid values (see inclusion criteria).

   (NUTRITIVE) INTERVENTION
   * Supplementation:

   A wash-out phase of at least 4 weeks, to eliminate all nutritional supplements taken prior to study, is followed by a 16 week long intervention phase. During this phase, the nutraceutical JP+ Omega Blend alone or in combination with an encapsulated fruit, vegetable and berry-juice concentrate (JP+Orchard, Garden and Vineyard blend; JP+OGV) will be supplemented. Participants allocated to the Ω2 group receive 2 capsules of JP+ Omega Blend/d, one capsule to be taken in the morning and one in the evening together with a meal. The intake of two capsules per day complies with the directions of use given on the label of the nutraceutical, which has been available on the market since 2016.

   Participants in the Ω4 group are instructed to consume 4 capsules of JP+ Omega Blend/d, two capsules along with the breakfast and two in the evening. In the Ω2+OGV group, participants receive 2 capsules of JP+® Omega Blend plus 2 capsules each of an encapsulated fruit, vegetable and berry-juice concentrate (JP+OGV) (total intake of 8 capsules/d; 4 capsules with the breakfast meal and 4 administered with the evening meal). The control group does not receive any supplementation. However, the subjects in this group are instructed not to change dietary habits during the 4 month long study period, similarly to the other intervention groups.

   All participants will be provided with a sufficient amount of supplements, according to their randomization group.

   Participants randomized into Ω2 receive 2 containers (with 60 capsules each) of the supplement at baseline and another 2 containers at the midpoint visit after 8 weeks. Ω4 participants receive twice the amount of the JP+Omega Blend capsules. Subjects in Ω2+OGV receive the same amount of JP+ Omega Blend capsules as Ω2 plus 2 containers each (containing 120 capsules) of JP+fruit, vegetable and berry juice concentrate.

   In total 2 backups will be retained for each intervention group and stored at room temperature. One full backup remains at the testing facility (Institute for Pathophysiology and Immunology), the second backup will be stored at Green Beat (Institute of Nutrient Research and Sport Nutrition). Thus, even in the case of the cancellation of a study visit (alternative visit scheduled within two weeks; elimination from the study after a longer period of absence from the visits), capsules should be available in sufficient amounts.

   Compliance: All participants will be asked to return the containers with the remaining capsules at the midpoint and endpoint visit. The capsules will be counted to determine the compliance of capsule intake.

   • Composition of the herbal omega-3 fatty acid nutraceutical

   Ingredients Amount per serving pro (2 capsules) Calories 15 kcal Total fat 1,5 g Proprietary blend of algal oil, pomegranate seed oil, sea buckthorn berry oil, raspberry seed oil, safflower seed oil, tomato seed oil 1354 mg

   Typically providing the following fatty acid profile:

   Total Omega Blend 925 mg Omega-3 375 mg DHA 175 mg EPA 100 mg ALA 50 mg Omega 5 + 7 Fettsäuren 250 mg Omega 6 + 9 Fettsäuren 300 mg Other Ingredients: Tapioca pullulan, silicon dioxide, orange oil, vanilla oil, rosemary oil.

   Ingredients: DHA- and EPA-enriched oil of the micro algae Schizochytrium sp. (with high oleic sunflower oil, antioxidant: rosemary extract, Tocopherol-rich extracs, ascorbylpalmitate), pomegranate seed oil 17 %, coating agent: pullulan; raspberry seed oil 11,5 %, sea buckthorn oil 9 %, release agent: silicon dioxide; high oleic safflower seed oil, tomatoe seed oil, orange oil, vanilla oil, antioxidant: rosemary extract.
   * Composition of the Juice Plus+ Orchard, Garden and Vineyard blend Juice Plus+® is an encapsulated, powdered juice concentrate derived from 36 different fruits, vegetables and berries including juice and pulp from concord grape, blueberry, cranberry, blackberry, bilberry, raspberry, redcurrant, blackcurrant, elderberry, green tea, ginger root, grape seed, artichoke leaf, cocoa, pomegranate, apple, orange, pineapple, cranberry, peach, acerola cherry, papaya, beet root, date, prune, carrot, parsley, beet, kale, broccoli, cabbage, tomato, spinach, sugar beet, garlic, as well as oat bran and rice bran. Six capsules (two of each Juice Plus+® OGV, respectively) of the nutraceutical provide 9.5 mg beta-carotene, 214 mg vitamin C, 60 mg vitamin E, 600 mcg folate and 63 kJ per day (= 6 capsules). The nutraceutical is distributed by the Juice Plus Company/NSA LLC, Collierville, TN, USA and manufactured for Europe by Natural Alternitives International (NAI), Manno, Switzerland.
   * Nutrition Subjects are instructed to implement a wash-out phase of any nutritional supplements and medication recently taken that could influence the outcome parameters of the study (especially omega-3 fatty acid supplements, plant extracts and concentrates). This phase should be implemented for at least 4 weeks of duration and will be standardized for nutrition intake of omega-3 fatty acid rich foods. Subjects are instructed to limit the intake of fish to maximal 1 portion/week, limit the intake of certain oils and nuts to maximal 1 Tbsp./d of rapeseed oil and 1 Tsp./d of linseed oil, hempseed oil, walnut oil; maximal 1 portion of nuts and seeds (25g)/d), as well as reduce the consumption if fruits and vegetables to maximal 3 portions/d (of which 2 portions may be vegetables).

   Before each of the fasted blood samples the participant's nutrition will be strictly standardized. Each of the subjects is instructed to protocol complete nutrition in the last 3 days before the baseline visit (and blood sample). Those protocols will be examined by a trained dietician and provide guidance for the participants. By this they can repeat the protocol and therefore reproduce the same nutritional intake in the days before the subsequent blood samples both at midpoint and endpoint visit.

   Dietary records developed by Green Beat are used, which have already been successfully established in different scientific studies. Additionally, these protocols collect information on physical activity, sleeping behaviour, as well as stress and well-being. All subjects receive a thorough instruction by a dietician on how to fill in the protocol.

   Summary of measures to standardize participant's nutrition:
   * max. 2 portions of fish/week
   * max. 3 portions of vegetables & fruit /d (of which max. 2 portions can be vegetables)
   * nuts and seeds: max. 1 portion (25g) / d
   * high quality, cold pressed oils: max. 1 Tbsp. rapeseed oil and 1 Tsp. per day of linseed oil, hempseed oil, walnut oil

   EVALUATION/STATISTICS Per protocol analyses will be performed with SPSS for Windows Software, Version 22.0. Data will be presented as mean ± SD. The randomisation of the subjects into the intervention groups will be considered during data analysis. Statistical significance is set at P < 0.05. The Shapiro-Wilk test will be used to determine normal distribution. Baseline characteristics (weight, age, gender, BMI etc.) of subjects will be determined by means of descriptive statistics and will be displayed graphically or in tables.

   Comparison of the mean values of baseline parameters among the 4 intervention groups will be done by analysis of variance, ANOVA. If data are normally distributed and variance homogeneity is fulfilled, student's t-test will be the main statistical test used to compare baseline and endpoint parameters in the respective group or to determine differences between baseline and midpoint, as well as midpoint and endpoint measurements. If it is not possible to use metrical data, non-parametric tests will be used (Wilcoxon rank sum test).

   One and two factorial repeated measures analysis of variance (ANOVA) are used to perform within and between group analysis for the factors "time" and "treatment", respectively. If the detected differences between the groups are significant, Tukey's post hoc test and Bonferroni correction will be used to determine the localization of the differences. In the case of the use of non-parametrical tests, Friedman Test (within group) and Kruskal Wallis test (between group) will be used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* 80 healthy men and women, 20-65 years
* suboptimal serum lipid values without medication
* triglycerides >140 mg/dl
* HDL Chol < 45 (m) or < 50 mg/dl (w)
* Non smokers
* BMI >20 and <35 kg/m2
* ω-3-fatty acid index (ω-3 index): rank 21 - 100 of the ranking or ω-3 index < 8%
* normal nutrition (omnivore diet)
* adherence to the 4-week long wash-out period

Exclusion criteria:

* all people not meeting the inclusion criterions
* hypertension (systolic blood pressure > 160mmHg, diastolic blood pressure >100 mmHg)
* Specific diets and nutritional habits (vegan, vegetarian, paleo, low-carb pregnancy)
* aversion to stop the intake of nutritional supplements and food, that could interfere with the study outcome
* over-consumption of fish (> 1 portion/week)
* linseed and walnut oil, whole linseeds and walnuts (>1 portion (25g)/day)
* with omega-3 fatty acids enriched "functional food
* intake of lipid-lowering, anti-inflammatory, blood pressure lowering medication and anticoagulants
* clinically relevant infectious disease
* acute and chronic inflammatory disease
* Diabetes mellitus type I and type II
* supplementation of antioxidants in all variations, omega-3 fatty acids, plant extracts/concentrates

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
Omega 3 index | 4 months
  Omega 3 index in erythrocytes is a valid parameter to estimate bioavailability of omega 3 fatty acids

SECONDARY OUTCOMES:
Change in lipid profile | 4 months
  Lipid metabolism may change over the time in a positive manner due to micronutrient intervention

OTHER OUTCOMES:
Micronutrient Absorption | 4 months
  Absorption of ß-carotene, tocopherols, vitamin A and vitamin C after 8 and 16 weeks of supplementation, measured via HPLC, proven by a UV detector, analysed by means of an internal standard method, evaluated by paired t-test, and assessed via SPSS 22.0

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Lamprecht, PhD,PhD, Study Chair — Green Beat and Medical University of Graz, Austria
Locations (2):
- Austria (2):
  - Institute of Pathophysiology and Immunology, Graz, Styria
  - Green Beat, Graz

IPD SHARING:
Plan to Share IPD: No